CLINICAL TRIAL: NCT06074549
Title: DynamX Bioadaptor Global Post-Market Registry: Clinical Trial of the Elixir Medical DynamX Coronary Bioadaptor System (Bio-RESTORE)
Brief Title: DynamX Bioadaptor Global Post-Market Registry: Clinical Trial of the Elixir Medical DynamX Coronary Bioadaptor System
Acronym: Bio-RESTORE
Status: Recruiting | Type: Observational
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ELX-CL-2002
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Open Label: DynamX Novolimus-eluting Coronary Bioadaptor System
  Interventions: Device: DynamX Novolimus-eluting Coronary Bioadaptor System

INTERVENTIONS:
Device: DynamX Novolimus-eluting Coronary Bioadaptor System — All patients will receive at least one DynamX Bioadaptor implant in a commercial setting in accordance with the product's Instructions for Use
  Other Names: DynamX Bioadaptor

SUMMARY:
The goal of this registry is to confirm the safety, and performance of the DynamX Coronary Bioadaptor System in patients with coronary artery disease.

DETAILED DESCRIPTION:
This registry will obtain additional safety, effectiveness, and performance data on the DynamX Coronary Bioadaptor System in the treatment of patients with ischemic heart disease due to de novo native coronary artery lesions in a real-world patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Patient understands the trial requirements and treatment procedures and provides informed consent
3. Patient indicated for PCI with stent implantation and receive at least one DynamX Bioadaptor implant in accordance with the product's Instructions for Use (IFU).

Exclusion Criteria:

1. Target Lesion(s) in the left main artery
2. Prior venous or arterial bypass grafts
3. In-stent restenosis
4. Patient is currently participating in another clinical trial with an investigational device or an investigational drug that has the potential to impact study results (e.g., anti-thrombotic or anti-platelet medications) that has not yet completed its primary endpoint
5. Patient is, in the opinion of the Investigator, unable to comply with the requirements of the study protocol or is unsuitable for the registry for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Percutaneous Coronary Intervention (PCI) who receive at least one DynamX Bioadaptor implant in a commercial setting in accordance with the product's Instructions for Use (IFU).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Device Oriented Clinical Endpoint | 12 Months
  Composite of Target Lesion Failure (TLF): cardiovascular death, target vessel myocardial infarction (TV-MI), or clinically indicated target lesion revascularization (CI-TLR), per ARC-2

SECONDARY OUTCOMES:
Clinical Device Success | In-Hospital, assessed up to 7 days after procedure
  Achievement of a final residual stenosis <30% by QCA or visual estimation, using the study device and without a device deficiency
Clinical Procedural Success | In-Hospital, assessed up to 7 days after procedure
  Achievement of a final residual stenosis <30% by QCA or visual estimation, using the study device, with or without any adjunctive devices, and without TLF
Device Oriented Clinical Endpoint | 30 days
  Composite of TLF: cardiovascular death, target vessel myocardial infarction (TV-MI), or clinically indicated target lesion revascularization (CI-TLR), per ARC-2
Patient Oriented Clinical Endpoint | 30 days and 12 months
  Composite of all-cause death, any stroke, any myocardial infarction (MI) (includes non-target vessel territory) and any revascularization.
Rate of target vessel failure (TVF) | 30 days and 12 months
  Composite of cardiovascular death, TV-MI, or target vessel revascularization (TVR).
Rate of all revascularization | 30 days and 12 months
  Target lesion, target vessel, non-target lesion, non-target vessel; clinically driven and non-clinically driven.
Rate of all MI | 30 days and 12 months
  Target and non-target vessel
Rate of all-cause death | 30 days and 12 months
  Cardiovascular, Non-Cardiovascular, Unknown
Composite of cardiovascular death, any myocardial infarction, and any revascularization | 30 days and 12 months
Rate of stroke | 30 days and 12 months
Rate of probable or definite stent thrombosis | 30 days and 12 months
Duration of DAPT | 30 days and 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- University Hospital St. Pölten, Pölten, Austria
- Curaçao Medical Center, Willemstad, Curacao
- Indonesia (4):
  - Heartology Cardiovascular Hospital, Jakarta
  - Jakarta Heart Center, Jakarta
  - Medistra Hospital, Jakarta
  - Siloam Hospitals, Jakarta
- Italy (3):
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Policlinico Tor Vergata, Rome
- Jordan (2):
  - Jordon Hospital, Amman
  - The Specialty Hospital, Amman
- King Fahad Armed Forces Hospital, Jeddah, Saudi Arabia
- Turkey (Türkiye) (2):
  - Istanbul Medipol Mega University Hospital, Istanbul
  - Memorial Bahçelievler Hospital, Istanbul
- Al Qassimi Hospital, Sharjah city, United Arab Emirates
- Vietnam (2):
  - Tam Duc Heart Hospital, Ho Chi Minh City
  - Kiến Giang General Hospital, Kiến Giang